CLINICAL TRIAL: NCT06494176
Title: Disseminable Evidence-Based Treatment for the Dental Office: Virtual Exposure Tools for Dental Fear - neVR Fear the Dentist
Brief Title: Virtual Reality Exposure for Dental Fear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s23-00772
Record Dates: First submitted 2024-05-16; First posted 2024-07-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Dental Fear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRET Intervention (Experimental)
  Interventions: Behavioral: neVR Fear the Dentist
- Active Control (No Intervention)

INTERVENTIONS:
Behavioral: neVR Fear the Dentist — neVR Fear the DentistTM comprises two major evidence-based interventions. First is a self-administered eHealth app for CBT/ psychoeducation with exposure therapy - delivered via a mobile tablet - that can be completed anywhere. Second is a 1-hr virtual reality exposure treatment (VRET).
  Arms: VRET Intervention

SUMMARY:
The purpose of this study is to compare an intervention for dental fear to the usual approach (i.e., whatever your dentist typically does to help you manage fear) in reducing patient fear and making dentist appointments more tolerable. The dental fear intervention (called neVR Fear the Dentist™) has two separate steps. Step 1 involves using a mobile app that is based on research-backed approaches to handling dental fear on your smartphone or device. Step 2 is a 1-hour self-administered virtual reality intervention to be completed in the dental office.

This is a randomized study. Participants will be randomized to either the intervention group or an active control.

Investigators hypothesize that participants in the intervention condition will show greater declines in self-reported dental fear and improved oral health-related quality of life during post-treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 13 years of age
2. Report dental fear of 4 or higher on a scale of 0-10 on the Gatchel dental fear item
3. Be able and willing to comply with study procedures
4. Provide a signed and dated informed consent form
5. Proficient in English because the intervention is in English
6. Have access to a smartphone or tablet
7. If self-referred, have a dental appointment already scheduled with their own dentist.
8. If self-referred, live in the NYC metro area or are willing to travel to the NYU College of Dentistry.
9. If self-referred, have access to an Oculus headset and live in the U.S.

Exclusion Criteria:

1. Uncorrected, severe, or profound hearing or visual impairment such as stereoscopy blindness or nystagmus
2. Diagnosed with any of the following psychiatric conditions: Posttraumatic Stress Disorder (PTSD) due to dental trauma, Major Neurocognitive Disorder (Dementia), Schizophrenia, or Intellectual Disability
3. Current diagnosis of a balance disorder, such as vertigo
4. Lifetime history of cybersickness
5. Previous history of epileptic seizures
6. A history of cardiac problems
7. Are in pain, require urgent care, or whose necessary treatment will be delayed by participating in the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in dental fear | Measure will be collected at baseline, immediately post-treatment, and 1-, 3-, and 6-months post treatment.
  Overall dental fear will be measured by the self-report Gatchel Dental Fear Item (Gatchel, 1987). This scale uses a one-item assessment of overall dental fear. Patients rate their dental fear on a scale of 0 = "None" to 10 = "High", with higher scores representing higher levels of fear.
Dental fear and anxiety | Measure will be collected at baseline, immediately post-treatment, and 1-, 3-, and 6-months post treatment.
  Dental fear and anxiety will also be measured using the Index of Dental Fear and Anxiety (IDAF; Armfield, 2010), an 8-item patient-report survey. Responses range from 1 = "Disagree" to 5 = "Strongly Agree." Total scores range from 5 to 40 with higher scores representing more dental anxiety/fear.
Anticipatory dental fear | Measure will be collected at baseline, immediately post-treatment, and 1-, 3-, and 6-months post treatment.
  Anticipatory dental fear will be measured via self-report using the Modified Dental Anxiety Scale (MDAS; Humphries et al., 1995), a 5-item scale. All items are rated on a 1-5 scale where 1 = "Not Anxious" and 5 = "Extremely Anxious," with total scores ranging from 5 to 25. Higher scores indicate higher dental anticipatory anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Heyman, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States